CLINICAL TRIAL: NCT06829355
Title: Efficacy and Safety Study of Thymalfasin in Combination with Targeted Immunotherapy (Regorafenib and Tislelizumab) in Patients with Advanced PMMR/MSS Colorectal Cancer Who Failed Standard of Care: a Multicenter, Open-label, Randomized, Controlled Clinical Study
Brief Title: "Thymalfasin Immunotherapy Study with Triple Regimen in Advanced MSS/pMMR Colorectal Cancer"
Acronym: THYMI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH-THYMIS; BFHHZML20240020 (Registry Identifier: Beijing Friendship Hospital, Capital Medical University)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: MCRC
Keywords: Thymalfasin; Regorafenib; Tislelizumab; mCRC; Combination; Immunotherapy; RCT
MeSH Terms: interventions — Thymalfasin; Trace amine-associated receptor 1; regorafenib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triple therapy group (Experimental): Subjects will receive Thymalfasin in combination with Regorafenib and Tislelizumab
  Interventions: Drug: Thymalfasin (Thymosin alpha 1, Ta1); Drug: Regorafenib (BAY 73-4506); Drug: Tislelizumab (BGB-A317)
- Double therapy group (Active Comparator): Subjects will receive Regorafenib and Tislelizumab
  Interventions: Drug: Regorafenib (BAY 73-4506); Drug: Tislelizumab (BGB-A317)

INTERVENTIONS:
Drug: Thymalfasin (Thymosin alpha 1, Ta1) — Thymalfasin: 4.8 mg, administered subcutaneously twice weekly.
  Arms: Triple therapy group
Drug: Regorafenib (BAY 73-4506) — Regorafenib: Start at 80 mg once daily, orally, taken at a fixed time for 2 consecutive weeks and then stopped for 1 week. If the patient tolerates it well, increase to 120 mg/d in Cycle 2.
Drug: Tislelizumab (BGB-A317) — Tislelizumab: 200 mg, iv.gtt, single infusion, 21 days as a cycle, Day 1.

SUMMARY:
This is a multicenter, open-label, prospective, randomized controlled Phase II clinical study. All eligible subjects will be randomly assigned in a 1:1 ratio to either the triple therapy group or the double therapy group.

Triple therapy group: Subjects will receive Thymalfasin in combination with Regorafenib and Tislelizumab until iCPD is achieved per iRECIST (progressive disease (PD) per iRECIST), or until an intolerable toxicity occurs; Double therapy group: Subjects will receive Regorafenib and Tislelizumab until iCPD is achieved per iRECIST (PD per iRECIST), or until an intolerable toxicity occurs.

DETAILED DESCRIPTION:
Assuming the following hypotheses:

H0: The mPFS of the test group minus the mPFS of the control group equals 0 H1: The mPFS of the test group minus the mPFS of the control group does not equal 0 Assuming an mPFS of 5.0 months for the test group and 1.8 months for the control group, with a two-sided alpha level of 0.05 and 80% power, at least 32 events need to be observed. Within a 9-month enrollment period and a total study duration of 15 months, 44 subjects need to be enrolled to achieve this. Considering an additional dropout rate of 15%, 26 subjects per group are required, totaling 52 subjects (using PASS 2023 Log-rank procedure).

Enrollment sites: Beijing Friendship Hospital, Capital Medical University, Peking Union Medical College Hospital, Peking University People's Hospital.

Allocation of enrollment across sites: Each site will compete for enrollment, with each site enrolling no less than 14 subjects.

1. Regorafenib: Start at 80 mg once daily, orally, taken at a fixed time for 2 consecutive weeks and then stopped for 1 week. If the patient tolerates it well, increase to 120 mg/d in Cycle 2.
2. Tislelizumab: 200 mg, iv.gtt, single infusion, 21 days as a cycle, Day 1.
3. Thymalfasin: 4.8 mg, administered subcutaneously twice weekly. Treatment will continue until disease progression or until an intolerable adverse reaction occurs that does not resolve despite dose modification.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign a written informed consent form (ICF) and able to understand and comply with the requirements of this study Male or female aged 18 to 75 Histologically or cytologically confirmed advanced or metastatic colorectal adenocarcinoma Mismatch repair (MMR) protein expression or microsatellite instability (MSI) testing showing pMMR/MSS ECOG score of 0 or 1 At least one measurable lesion per iRECIST Expected survival of ≥ 3 months Disease progression or intolerance after at least second-line standard systemic therapy

Normal major organ function and hematological parameters (within 14 days prior to randomization):

Hematology tests must meet the following criteria:

WBCs≥2.0×10^9/L NEUT≥1.5×10^9/L Hb≥90g/L (9.0g/dL); PLT ≥100×10^9/L;

Biochemistry tests must meet the following criteria:

TBIL ≤ 1.5 × upper limit of normal (ULN); Without liver metastases, ALT or AST ≤ 3.0 ULN; with liver metastases, ALT or AST ≤ 5 ULN; Serum albumin level ≥ 30 g/L Serum Cr ≤ 1.5 ULN, with an endogenous creatinine clearance (CrCl) > 40 mL/min (using Cockcroft-Gault formula) For females: CrCl =((140-Age）×Weight（kg）× 0.85)/(72 × Cr (mg/dL)) For males: CrCl =((140-Age）×Weight（kg）× 1.00)/(72 × Cr (mg/dL)) Urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein must be < 1 g Prothrombin time or activated partial thromboplastin time and international normalized ratio ≤ 1.5 × ULN Able to swallow and absorb oral medication Females of childbearing potential must use appropriate contraceptive methods during the study and for 6 months after the last dose of the study drug. For males, they should be surgically sterilized or agree to use appropriate contraceptive methods during the study and for 6 months after the last dose of the study drug.

Exclusion Criteria:

* 1. Previous treatment with Regorafenib, PD-1, PD-L1, or CTLA-4 inhibitors, or any form of immunotherapy; 2. Treatment with related drugs or medical technology affecting immunity within 6 months prior to the first dose of the study drug (including but not limited to: thymopentin, interferon, tumor vaccines, CAR-T therapy, etc.); 3. Receiving any study drug, radiotherapy, or major surgery within 28 days prior to the first dose of the study drug; 4. Receiving any anti-tumor treatment (chemotherapy, targeted therapy, etc.) within 3 weeks prior to the first dose of the study drug; 5. Presence of symptomatic central nervous system (CNS) metastases or CNS metastases requiring local CNS-directed therapy (such as radiotherapy or surgery). Exceptions include those previously treated and stable for ≥ 2 months and who have stopped systemic treatment for more than 4 weeks prior to the first dose of the study drug; 6. Known allergy or intolerance to any of the study drugs or their components; 7. Pregnant or lactating females; 8. History of other malignant tumors within the past 5 years (excluding carcinoma in situ or basal cell or squamous cell skin cancer; subjects with other malignant tumors who have been cured for at least 5 years are eligible); 9. Symptomatic congestive heart failure (NYHA Class II-IV), symptomatic or uncontrolled arrhythmias; 10. Poorly controlled hypertension, defined as systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite best medical treatment; 11. Unstable angina (angina symptoms at rest), new onset angina (within the past 3 months), or myocardial infarction within 6 months prior to the first dose of the study drug; 12. Major thrombotic or bleeding events within 6 months prior to randomization (including hemoptysis, gastrointestinal bleeding, hematemesis, central nervous system (CNS) bleeding, severe epistaxis or vaginal bleeding, cerebral infarction, transient ischemic attack, or uncontrolled coronary heart disease). Or requiring lifelong oral anticoagulant therapy; 13. With active, known, or suspected autoimmune diseases; 14. Receiving immunosuppressive agents within 4 weeks prior to the first dose of the study drug, excluding topical glucocorticoids or physiological doses of systemic glucocorticoids administered by nasal, inhalation, or other routes (i.e., no more than 10 mg prednisolone per day or equivalent dosage of other glucocorticoids); 15. Diagnosed with immunodeficiency or on chronic systemic steroid therapy (at a dose in excess of 10 mg prednisone equivalent per day) or any other form of immunosuppressive therapy; 16. History of interstitial lung disease; 17. Active tuberculosis requiring anti-tuberculosis treatment or treatment for tuberculosis within 1 year prior to the first dose of the study drug; 18. Acute or chronic active hepatitis B or hepatitis C; 19. Known history of human immunodeficiency virus (HIV) or syphilis infection; 20. Other active or severe infections requiring systemic antibacterial, antifungal, or antiviral treatment within 4 weeks prior to the first dose of the study drug; 21. Unresolved clinical toxicity ≥ Grade 2 (NCI-CTCAE, v5.0) due to prior anti-tumor treatment, excluding alopecia or non-clinically significant laboratory abnormalities; 22. Intestinal obstruction, gastrointestinal perforation, Crohn's disease, ulcerative colitis, abdominal abscess, chronic diarrhea, or fistula disease within 6 months prior to enrollment; 23. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B or more severe cirrhosis; 24. Vaccination with live vaccines within 30 days prior to planned initiation of the study drug (seasonal influenza vaccines without live virus are permitted); 25. History of alcohol abuse or drug abuse; 26. Other acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that the investigator believes would make the use of the study drug unfavorable or affect the interpretation of AEs, or, in the investigator's judgment, would result in inadequate compliance during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-02-11 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 48 WEEKS
  Time from day of randomization to the date of documented tumor progression or death due to any cause

SECONDARY OUTCOMES:
18-week PFS rate | 18 weeks
  Proportion of patients without disease progression or death at 18 weeks after starting the study treatment.
Objective response rate (ORR) | 48 WEEKS
  Proportion of patients with tumor size reduction of a predefined amount and maintaining for a certain time period, ORR = CR + PR
Disease control rate (DCR) | 48 WEEKS
  Proportion of patients with tumor control with tumor size reduction of a predefined amount and maintaining for a certain time period, DCR = CR + PR + SD
Overall survival (OS) | 3 Years
  Time from day of randomization to death due to any cause.
1-year OS rate | 48 WEEKS
  Proportion of patients alive at 1 year after starting the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Professor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided